CLINICAL TRIAL: NCT01362816
Title: The European Palliative Care Cancer Symptom Study (EPCCS). A Prospective Data Collection
Brief Title: The European Palliative Care Cancer Symptom Study (EPCCS)
Acronym: EPCCS
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Rigshospitalet, Denmark (Other); Oslo University Hospital (Other); Medical University of Graz (Other); University of Navarra (Other); Hospital Universitario La Paz (Other); Cantonal Hospital of St. Gallen (Other); Institut Català d'Oncologia (Other); University of Alberta (Other); Flinders University (Other); University Hospital, Ghent (Other); The Cleveland Clinic (Other); Hospital de San Lázaro (Unknown); Haukeland University Hospital (Other); Kantonsspital Graubünden (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); University of Edinburgh (Other); Leeds Cancer Centre at St. James's University Hospital (Other); Turku University Hospital (Other Government); St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/2945-3
Record Dates: First submitted 2011-05-27; First posted 2011-05-30 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Palliative care cancer patients: Inclusion criteria are:
  Patient has a cancer diagnosis (radiological, histological, cytological or operative evidence), local, loco-regional or metastatic disease, defined as a palliative care patient; enrolled in a palliative care programme, age 18 years or older, able to provide written informed consent, able to complete the data collection tool, preferably without help, available for follow up registration

SUMMARY:
The rising incidence of cancer and the rapidly increasing number of people living longer with incurable disease, accentuates the need for optimal symptom management throughout the disease trajectory. Thanks to the medical and technological development, and the increased interest in palliative care research, palliative medicine has gradually become more evidence based. Patients with advanced cancer experience multiple symptoms at the time with fluctuating intensity and severity. Pain, fatigue, nausea/vomiting, dyspnea, loss of appetite and depression are among the most common and experienced by more than 50%. However, the prevalence rates of these symptoms vary considerably across studies, with a range from 35 to 90 % for pain as an example. These differences may in part be explained by different assessment tools, study methods and design and population characteristics. There is also lack of agreed-upon, common criteria to describe the main characteristics of a palliative care cancer population and few standardized tools for assessment and classification of symptoms exist. These shortcomings limit the possibility to design randomized controlled treatment trials in palliative care; the optimal way to improve clinical symptom management. To do this, a better understanding of how symptoms evolve and how they should be assessed and classified throughout the palliative care disease trajectory is important, supplemented with registrations of the treatment provided. The primary aim of this international research project the European Palliative Care Cancer Symptom study (EPCCS) is to extend the knowledge about and gain new insight in the prevalence and development of the most frequent cancer related symptoms during the course of disease, in a large sample of palliative care cancer patients. The clinical usefulness of the new assessment and classification system developed by the European Palliative Care Research Collaborative (EPCRC) / European Association for Palliative Care Research Network (EAPC RN) will be examined and data on the organization and delivery of palliative care at participating centers will be collected. The project also aims to further develop and consolidate international research collaboration through the European Palliative Care Research Centre (PRC). Taken together, these efforts will increase the understanding of the palliative disease trajectory and provide necessary knowledge and structure for future randomized controlled trials (RCTs)

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a cancer diagnosis (radiological, histological, cytological or operative evidence)
2. Local, loco-regional or metastatic disease
3. Defined as a palliative care patient; enrolled in a palliative care programme
4. Age 18 years or older
5. Able to provide written informed consent
6. Able to complete the data collection tool, preferably without help
7. Available for follow up registration

Exclusion Criteria:

1. Patients receiving anti-cancer treatment with a curative intent
2. Patients who are unable to complete the registration due to language problems or severe physical problems
3. Patients who have psychotic disorders or obvious cognitive impairment
4. Patients who cannot come for regular follow-up visits, due to geographical or social reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The popuation consists of patients with incurable cancers who are enrolled in a palliative care programme. They will be identified upon referral for non-curative cancer treatment/palliative care to the centre, department, out-patient clinic, daycare centre, hospice, or home-based care, depending on the palliaitve care organization model at the participating centres. Patients will be followed every 4 weeks (3-5) for at least 6 months, or until death
Sampling Method: Non-Probability Sample
Enrollment: 1739 (Actual)
Dates: Start 2011-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
change in cancer symptoms | up to 6 months
  assessment and classification system developed by the European Palliative Care Research Collaborative (EPCRC) / European Association for Palliative Care Research Network (EAPC RN)

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, Prof MD, Principal Investigator — Norwegian University of Science and Technology; Marianne J Hjermstad, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Ekstrom M, Johnson MJ, Schioler L, Kaasa S, Hjermstad MJ, Currow DC. Who experiences higher and increasing breathlessness in advanced cancer? The longitudinal EPCCS Study. Support Care Cancer. 2016 Sep;24(9):3803-11. doi: 10.1007/s00520-016-3207-1. Epub 2016 Apr 9. PMID 27061408
- [Derived] Ekstrom MP, Palmqvist S, Currow DC, Sjogren P, Kurita GP, Jakobsen G, Kaasa S, Hjermstad M. Mild to Moderate Cognitive Impairment Does Not Affect the Ability to Self-Report Important Symptoms in Patients With Cancer: A Prospective Longitudinal Multinational Study (EPCCS). J Pain Symptom Manage. 2020 Aug;60(2):346-354.e2. doi: 10.1016/j.jpainsymman.2020.03.007. Epub 2020 Mar 14. PMID 32179133
- [Derived] Vagnildhaug OM, Brunelli C, Hjermstad MJ, Strasser F, Baracos V, Wilcock A, Nabal M, Kaasa S, Laird B, Solheim TS. A prospective study examining cachexia predictors in patients with incurable cancer. BMC Palliat Care. 2019 Jun 4;18(1):46. doi: 10.1186/s12904-019-0429-2. PMID 31164115
- [Derived] Boland JW, Allgar V, Boland EG, Kaasa S, Hjermstad MJ, Johnson MJ. Predictors and trajectory of performance status in patients with advanced cancer: A secondary data analysis of the international European Palliative Care Cancer Symptom study. Palliat Med. 2019 Feb;33(2):206-212. doi: 10.1177/0269216318811011. Epub 2018 Nov 8. PMID 30404572
- [Derived] Habberstad R, Hjermstad MJ, Brunelli C, Kaasa S, Bennett MI, Pardon K, Klepstad P. Which factors can aid clinicians to identify a risk of pain during the following month in patients with bone metastases? A longitudinal analyses. Support Care Cancer. 2019 Apr;27(4):1335-1343. doi: 10.1007/s00520-018-4405-9. Epub 2018 Aug 13. PMID 30105665
- [Derived] Paque K, Elseviers M, Vander Stichele R, Pardon K, Hjermstad MJ, Kaasa S, Dilles T, De Laat M, Van Belle S, Christiaens T, Deliens L. Changes in medication use in a cohort of patients with advanced cancer: The international multicentre prospective European Palliative Care Cancer Symptom study. Palliat Med. 2018 Apr;32(4):775-785. doi: 10.1177/0269216317746843. Epub 2017 Dec 15. PMID 29243546
- [Derived] Hjermstad MJ, Aass N, Aielli F, Bennett M, Brunelli C, Caraceni A, Cavanna L, Fassbender K, Feio M, Haugen DF, Jakobsen G, Laird B, Lohre ET, Martinez M, Nabal M, Noguera-Tejedor A, Pardon K, Pigni A, Piva L, Porta-Sales J, Rizzi F, Rondini E, Sjogren P, Strasser F, Turriziani A, Kaasa S; European Palliative Care Cancer Symptom study (EPCCS). Characteristics of the case mix, organisation and delivery in cancer palliative care: a challenge for good-quality research. BMJ Support Palliat Care. 2018 Dec;8(4):456-467. doi: 10.1136/bmjspcare-2015-000997. Epub 2016 May 31. PMID 27246166